CLINICAL TRIAL: NCT05258071
Title: A Randomised, Placebo-controlled, Multicentre Phase IIb Study Evaluating the Efficacy of Pirepemat on Falls Frequency in Patients with Parkinson's Disease
Brief Title: A Clinical Study Evaluating Efficacy of Pirepemat on Falls Frequency in Patients with Parkinson's Disease (PD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Integrative Research Laboratories AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRL752C003
Record Dates: First submitted 2022-02-10; First posted 2022-02-28 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Frequent fallers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pirepemat dose 1 (Experimental): Pirepemat tablets, dose 1 (mg), 2 tablets t.i.d. for 84 days.
  Interventions: Drug: Pirepemat
- Pirepemat dose 2 (Experimental): Pirepemat tablets, dose 2 (mg), 2 tablets t.i.d. for 84 days.
  Interventions: Drug: Pirepemat
- Placebo (Placebo Comparator): Placebo tablets, 2 tablets t.i.d. for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirepemat — Oral use
  Other Names: IRL752
  Arms: Pirepemat dose 1; Pirepemat dose 2
Drug: Placebo — Oral use
  Arms: Placebo

SUMMARY:
This is a Phase 2b study investigating the efficacy and safety of pirepemat as adjunct therapy on falls frequency in patients with Parkinson disease. Pirepemat is taken for 84 days.

DETAILED DESCRIPTION:
At the screening visit consenting patients will be screened for eligibility according to study specific inclusion/exclusion criteria within 6 weeks before start of Investigational Medicinal Product (IMP) administration. Patients will be asked to complete a fall diary for at least 4 consecutive weeks during the screening period and to be eligible for randomization, the patient should have experienced at least 2 falls during the 4 weeks preceding the baseline visit.

At the baseline visit, patients will be randomized to receive one of two doses of Pirepemat (dose 1 or dose 2) or placebo t.i.d. (1:1:1). Dosing will start with half the dose for the first week of treatment and then continue with full dose until Week 11. Dosing will be de-escalated according to pre-specified schedule during the last week of study treatment, ending with the last dose on Day 84.

The treatment allocation will be double-blind, i.e. it will not be disclosed to the patients, the site staff or the Sponsor.

During the treatment period, patients will capture falls at home using a fall diary and changes in cognitive, postural, motor and mental functions will be assessed using the Montreal Cognitive Assessment (MoCA), Movement Disorder Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS), Neuropsychiatric Inventory (NPI) (Apathy/Indifference part), Single Leg Stance Test, Tandem walking test, and Clinician's Global Impression of Severity (CGI-S) and Improvement (CGI-I).

Blood samples for pharmacokinetic (PK) analysis will be collected at visit 5 (week 6) and visit 8 (week 11).

Following the last IMP dose, a safety follow-up period (including laboratory assessments at 3 instances) of approximately 1 month will take place.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 55-85 years of age, inclusive.
2. Diagnosis of idiopathic Parkinson's disease, according to the UK Parkinson's disease Society Brain Bank criteria.
3. Montreal Cognitive Assessment (MoCA) score of ≥10 and <26 at screening.
4. A modified Hoehn & Yahr score of ≥2.5 in "on".
5. Having experienced recurrent falls during the past 3 months (based on interview with the patient and/or caregiver) and at least 2 falls during the past 4 weeks before baseline.
6. On a stable regimen of anti-Parkinson's medications for at least 30 days prior to baseline, and willing to continue the same doses and regimens during study participation.
7. Able to cooperate and participate in study related procedures. This includes the ability to accurately complete a fall diary. The fall diary may also be completed by a responsible caregiver. For patients meeting DSM-IV TR criteria for Parkinson's disease dementia, the fall diary should be completed by the caregiver.
8. Availability of a responsible caregiver at least five days per week at least 2 hours per day. For patients meeting DSM-IV TR criteria for Parkinson's disease dementia, availability of a responsible live-in caregiver is required.
9. Female patients must be of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal females defined as 12 months of amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulation hormone (FSH) 25-140 IE/L and oestradiol <200 pmol/L is confirmatory]).
10. Fertile male patients must be willing to use condom and refrain from donating sperm during the study and until 3 months after last dosing of IMP and ensure that their fertile female partners are using contraceptive methods to prevent pregnancy .
11. Written informed consent for participation in the study given by the patient and the responsible caregiver.

Exclusion Criteria:

1. Any of the following potential hepatic conditions:

   1. known history of alcohol abuse, chronic liver or biliary disease, with the exception of Gilbert's syndrome
   2. total bilirubin greater than the upper limit of the normal range (unless associated with isolated instances of suspected Gilbert's syndrome)
   3. alkaline phosphatase (ALP) greater than 1.5 times the upper limit of the normal range
   4. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2 times the upper limit of the normal range
   5. history of repeated unexplained upper right quadrant abdominal pain and/or nausea, or jaundice
2. A positive Hepatitis B surface antigen or a positive Hepatitis C antibody result.
3. A score of 5 (wheelchair bound or bedridden) in the "on"-state on the modified Hoehn & Yahr scale.
4. Uncontrolled symptomatic orthostatic hypotension.
5. Clinically significant polyneuropathy.
6. Weight <55 kg at Screening.
7. Patients with current or past treatment with deep brain stimulation (DBS) or patients with previous history of stereotaxic brain surgery for PD.
8. A current diagnosis of any primary neurodegenerative disorder other than idiopathic PD.
9. A current diagnosis of any treatable dementia (hypothyroidism, syphilis, vitamin B12 or folate deficiency) that is verified by the investigator to be the cause of dementia.
10. A current diagnosis of a major depressive episode according to DSM-IV criteria.
11. Patient has delirium.
12. Any history of a heart condition, including prolonged QTc (>450 ms for males and > 470 ms for females, QTcF and/or QTcB), cardiac arrhythmias, any repolarisation deficits or any other clinically significant abnormal ECG as judged by the Investigator.
13. Severe or ongoing unstable medical condition including a history of poorly controlled diabetes; obesity associated with metabolic syndrome; uncontrolled hypertension; cerebrovascular disease, or any form of clinically significant cardiac disease; renal failure, history of abnormal renal function.
14. History of seizures within two years of screening.
15. History of cancer within five years prior to screening, with the following exceptions: adequately treated non-melanomatous skin cancers, localised bladder cancer, non-metastatic prostate cancer or in situ cervical cancer.
16. History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to pirepemat.
17. Creatinine clearance <30 mL/min (calculated according to the Cockroft-Gault formula).
18. Treatment with Warfarin within three months before study treatment.
19. Treatment with Amantadine within 6 weeks before study treatment.
20. Treatment with Selegiline within 6 weeks before study treatment.
21. Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment with less than three months between administration of last dose and first dose of IMP in this study.
22. Current or history of drugs of abuse according to DSM-IV criteria.
23. Any planned major surgery within the duration of the study.
24. Any other condition or symptoms preventing the patient from entering the study, according to the Investigator's judgement.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Change in falls frequency with Pirepemat compared to placebo as assessed with fall diary from baseline period (4 weeks prior to randomization) to the end of treatment. | Baseline to end of treatment (week 12)
  Falls being recorded using a paper fall diary (Patient Reported Outcome, PRO)

SECONDARY OUTCOMES:
Change in the total score of MDS-UPDRS part 2 (M-EDL) from baseline to end of full dose treatment (with pirepemat compared to placebo). | Baseline to end of full dose treatment (week 11)
  The total scoring range is 0-52, where a higher score indicates more severe impact on Motor Aspects of Experiences of Daily Living (M-EDL).
Change in total score (Frequency*Severity) of NPI Item G (Apathy/Indifference) from baseline to end of full dose treatment (with pirepemat compared to placebo). | Baseline to end of full dose treatment (week 11)
  The total scoring range is 1-12, where a higher score indicates a higher degree of apathy/indifference.
Change in Caregiver distress of NPI Item G (Apathy/Indifference) from baseline to end of full dose treatment (with pirepemat compared to placebo). | Baseline to end of full dose treatment (week 11)
  The total scoring range is 0-5, where a higher score indicates a more severe caregiver distress.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Tedroff, Study Director — Integrative Research Laboratories AB
Locations (37):
- France (5):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Hopital de la Timone, Marseille
  - Hôpital Laennec - Centre d'investigation clinique de Neurologie, Nantes
  - CHU Charles Nicolle, Rouen
  - CHU Toulouse - Hôpital Purpan, Toulouse
- Germany (10):
  - Charite Universitatsmedizin Berlin - Klinik fuer neurologie mit experimenteller neurologie, Berlin
  - Praxis Dr.med. Christian Oehlwein Facharzt für Neurologie und Psychiatrie, Gera
  - Universitätsmedizin Göttingen - Klinik für Neurologie, Göttingen
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Universitaetsklinikum Leipzig - Klinik und Poliklinik fuer Neurologie, Leipzig
  - Philipps-Universitaet Marburg, Marburg
  - Kliniken Kreis Muehldorf a. Inn, Mühldorf
  - Universitysklinikum Münster - Klinik für neuroligie, Münster
  - Klinische Forschung Schwerin GmbH, Schwerin
  - RKU - Universitäts- und Rehabilitationskliniken Ulm Klinik für Neurologie, Ulm
- Radboud Universitair Medisch Centrum (Radboudumc), Nijmegen, Netherlands
- Poland (11):
  - Silmedic sp. z o.o, Katowice
  - Diamond Clinic sp. z o.o., Krakow
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - Pratia MCM Krakow, Krakow
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Instytut Zdrowia, Oświęcim
  - Centrum Medyczne HCP SP Z OO, Poznan
  - Neuro-Care Clinic, Siemianowice Śląskie
  - RCMed, Sochaczew
  - Centrum Medyczne NeuroProtect, Warsaw
  - Singua Sp. z o.o., Warsaw
- Spain (7):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Infanta Sofia, Madrid
  - Hospital Universitario del Henares, Madrid
  - Clinica Universitaria de Navarra, Pamplona
- Sweden (3):
  - Institute of Neuroscience and Physiology, Gothenburg
  - Skane University Hospital - Division of Neurology, Lund
  - Karolinska Universitetssjukhuset - Neurologiska kliniken, Stockholm